CLINICAL TRIAL: NCT03372317
Title: Tau Positron Emission Tomography (PET) in Imaging and Cognition
Brief Title: Tau PET in Imaging and Cognition: Healthy Adults From 55-90
Status: Recruiting | Type: Observational
Sponsor: Yaakov Stern (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Yaakov Stern, Professor of Neuropsychology, Columbia University
Organization: Columbia University (Other)
Other Study IDs: AAAR6959; 2RF1AG038465-06 (NIH)
Record Dates: First submitted 2017-12-08; First posted 2017-12-13 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Mild Cognitive Impairment; Aging
Keywords: Tau; MK-6240; Cognition
MeSH Terms: conditions — Cognitive Dysfunction; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma, serum and cells will be retained
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Non-demented elders: Participants aged 55-90 that are cognitively normal or have mild cognitive impairment will receive 18F-MK-6240 to identify the presence of tau protein in the brain.
  Interventions: Drug: 18F-MK-6240

INTERVENTIONS:
Drug: 18F-MK-6240 — Results of the 18F-MK-6240 PET scan will be correlated with other observations.
  Other Names: 6-[18F]Fluoro-3-(1H-pyrrolo[2,3-c]pyridin-1-yl)isoquinolin-5-amine

SUMMARY:
The investigators aim to use the new PET radioligand, 18F-MK-6240, to detect tau pathology in cognitive healthy and mild cognitive impairment (MCI) elders. The investigators will then examine the interactions between differential tau burden and performance on cognitive tasks, functional magnetic resonance imaging (fMRI) neural activation patterns, and other cognitive and behavioral measures. By investigating these relationships, the investigators hope to understand the cognitive and behavioral outcomes of tau deposition found in specific brain regions in cognitively normal/mildly cognitively impaired adults. Furthermore, the study aims to examine how the presence of tau may contribute to the risk of subsequent cognitive decline, neurodegeneration, and dementia.

DETAILED DESCRIPTION:
Many cognitively healthy older adults have, upon post mortem evaluations, been found to have varying amounts of neurofibrillary tangles (tau) and beta-amyloid plaque deposits, which are the hallmark brain pathologies known to be associated with Alzheimer's disease and various other dementias. While some with these pathologies may not clinically express cognitive decline or dementia in their lifetime, human post-mortem studies suggest that increasing neurofibrillary tangle density correlates with neurodegeneration and cognitive impairment.

Imaging tauopathy in-vivo provides an opportunity to examine neurocognitive correlates of differential levels of tauopathy in the brain, allowing to further qualify pre-clinical states of cognitive impairment. The investigators aim to investigate possible protective mechanisms, such as cognitive reserve, that may modulate the relationship between tauopathy and cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Aged 55-90
* Previously received an amyloid PET scan
* Residing near Columbia University Medical Center
* Must be willing and able to participate

Exclusion Criteria:

* Have a contraindication to PET (e.g, metallic implants, pacemaker, claustrophobia, or cannot lie flat for one hour)
* Pregnancy
* Lactating Women
* Current, past, or anticipated exposure to radiation
* Significant active physical illness

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects, 55-90 years old that previously received an amyloid PET scan
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Total number of individuals with tau present | Up to 5 years
  Based on the scans, the total number of subjects with identifiable tau in their scans will be measured.
Cognition | Up to 5 years
  Relation of Tau PET to measures of cognition such as memory and reasoning
Functional imaging (fMRI) | Up to 5 years
  Relation of Tau PET to imaging acquired during task performance

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Stern, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data could be shared based on NIH regulations
Time Frame: Study data will be available within 1 year
Access Criteria: We will be sharing de-identified data with a consortium that is aggregating studies that have employed tau PET tracers